CLINICAL TRIAL: NCT01812720
Title: A Phase 2 Trial of Carfilzomib Consolidation After Autologous Stem Cell Transplantation for Multiple Myeloma(CARAMEL 2)
Brief Title: Carfilzomib and Dexamethasone in Treating Patients With Multiple Myeloma Who Previously Underwent a Stem Cell Transplant
Acronym: CARAMEL 2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1287; NCI-2013-00492 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-005975; MC1287 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-01

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (carfilzomib, dexamethasone) (Experimental): Patients receive carfilzomib IV over 30 minutes and dexamethasone PO on days 1, 2, 15, and 16. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carfilzomib; Drug: dexamethasone; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well carfilzomib and dexamethasone work in treating patients with multiple myeloma who previously underwent a stem cell transplant. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunosuppressive therapy, such as dexamethasone, may improve bone marrow function and increase blood cell counts. Giving carfilzomib together with dexamethasone may be an effective treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the complete response (CR) rate with carfilzomib and dexamethasone consolidation following an upfront single stem cell transplant (SCT).

SECONDARY OBJECTIVES:

I. To assess the toxicity of carfilzomib and dexamethasone when used as consolidation therapy in patients post SCT.

II. To determine the progression free rate at 1 and 2 years post SCT. III. To evaluate progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To determine the proportion of patients achieving a minimal residual disease (MRD) negative status.

II. To assess the HevyLite assay prior to and during treatment.

OUTLINE:

Patients receive carfilzomib intravenously (IV) over 30 minutes and dexamethasone orally (PO) on days 1, 2, 15, and 16. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 3 years and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine =< 3 mg/dL
* Absolute neutrophil count >= 1,000/uL
* Platelet count >= 75,000/uL
* Hemoglobin >= 8.0 g/dL
* Previous diagnosis of symptomatic multiple myeloma (MM)
* Received single autologous stem cell transplantation 60-120 days prior to registration
* Received the autologous SCT =< 12 months of their diagnosis of myeloma to be eligible for the study
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Recovered from toxicity of previous chemotherapy (excludes grade 1 neurotoxicity and hematological toxicity)
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care
* Negative pregnancy test performed =< 7 days prior to registration, for women of childbearing potential only
* Willingness to return to one of the enrolling institutions for follow-up (during the active monitoring phase of the study); NOTE: during the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Measurable disease of multiple myeloma at the time of baseline values for disease assessment as defined by at least one of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * NOTE: for patients with no relapse prior to transplant, measurable disease at the time of diagnosis
  * NOTE: for patients who have had a disease relapse prior to transplant, measurable disease at the time of the most recent relapse immediately prior to transplant; NOTE: if the patient had treatment for the relapsed disease prior to transplant, the patient must have measurable disease at the time of relapse prior to this therapy
* Willing to provide bone marrow and blood samples for correlative research purposes

Exclusion Criteria:

* Prior allogeneic bone marrow/peripheral blood stem cell transplant
* Evidence of disease progression post SCT at the time of consideration for the study enrollment
* Myocardial infarction =< 6 months prior to registration
* New York Heart Association (NYHA) class III or IV heart failure
* Uncontrolled angina
* Severe uncontrolled ventricular arrhythmias
* Electrocardiographic (ECG) evidence of acute ischemia or active conduction system abnormalities; NOTE: prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant
* Seroreactivity for human immunodeficiency virus (HIV), human T-cell lymphotrophic virus (HTLV) I or II, hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Other active malignancy requiring therapy; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* Pregnant women or women of reproductive capability who are unwilling to use effective contraception
* Nursing women
* Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 28 days after stopping treatment
* Other co-morbidity, which would interfere with patient's ability to participate in the trial, e.g. uncontrolled infection, uncompensated lung disease
* Concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Known allergies to any of the components of the investigational treatment regimen or required ancillary treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Rate of complete response | Up to 5 years
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Overall survival | Time from registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Progression-free survival | Time from registration to progression or death due to any cause, assessed up to 5 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time to progression post SCT | Time from SCT to the earliest day with documentation of disease progression, assessed at 1 year post-SCT
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time to progression post SCT | Time from SCT to the earliest day with documentation of disease progression, assessed at 2 years post-SCT
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Maximum grade for each type of adverse event | Up to 30 days after last day of treatment
  Frequency tables will be reviewed to determine adverse event patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri